CLINICAL TRIAL: NCT05902676
Title: The Effects Of Anticholinergic Burden On Daily Living Activities In Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, hasan oztin, Head of Geriatrics, Izmir Ataturk Training and Research Hospital
Other Study IDs: 301-16/1648-946
Record Dates: First submitted 2023-05-22; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Anticholinergic Syndrome; Anticholinergic Adverse Reaction; Antispasmodic Adverse Reaction; Antiarrhythmic Drug Adverse Reaction; Antiparkinsonism Drugs Causing Adverse Effects in Therapeutic Use; Psychotropic Agents Causing Adverse Effects in Therapeutic Use
Keywords: anticholinergic burden; daily living activities; geriatrics
MeSH Terms: conditions — Anticholinergic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- no anticholinergic burden: Patients with a score of 0 were considered to have not used anticholinergic medications. Short-term use of medications, daily dosages of medications, and topical, ophthalmic, otologic, or inhalation medications were excluded from scoring.
- anticholinergic burden: Patients with a score of 1 or higher were considered to have used anticholinergic medication. Short-term use of medications, daily dosages of medications, and topical, ophthalmic, otologic, or inhalation medications were excluded from scoring.

SUMMARY:
The anticholinergic burden was calculated based on the medications that the patients had used for more than 10 days. Short-term medications used by patients were not evaluated. Among all the medications used by the patients, those with anticholinergic effects were scored according to the scale, and the total anticholinergic burden was calculated by adding them up. Those who had no anticholinergic score were considered to have no anticholinergic burden.

The study cohort will be stratified into two cohorts, distinguished by the presence or absence of anticholinergic burden. To evaluate the impact of anticholinergic burden on daily living activities and instrumental ADL, the groups will be compared with respect to hand grip strength and walking speed.In this study, the anticholinergic burden will be calculated based on medications used by the patients for more than 10 days, excluding short-term medications. Each medication with anticholinergic effects will be assigned a score according to a scale, and the total anticholinergic burden will be determined by summing up the scores. Patients without any anticholinergic score will be classified as having no anticholinergic burden.

The study cohort will be divided into two groups based on the presence or absence of anticholinergic burden. To assess the impact of anticholinergic burden on daily living activities (ADLs) and instrumental ADLs, the groups will be compared in terms of hand grip strength and walking speed.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years old
* Patients without a diagnosis of dementia and with MMSE>24
* Patients who can communicate (without hearing or visual problems)
* Those who give written consent to participate in the study

Exclusion Criteria:

* Patients with a diagnosis of dementia at their initial visit,
* Bedridden patients (those with visual impairments)
* Patients with walking difficulties (due to pain, prostheses, visual problems, etc.), vitamin D deficiency (10) (20ng/dl>) or those who use assistive devices (walker, cane, etc.) or those with sequelae of cerebrovascular events or hip fractures.
* Patients with a diagnosis of delirium,
* Those who underwent major surgery in the last 6 months,
* Those who experienced cardiac or cerebrovascular events during the follow-up period,
* Patients with infectious diseases,
* Those who did not sign or withdrew their consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A prospective case-control study was designed, and 180 patients over 65 years of age who applied to the geriatrics outpatient clinic without a diagnosis of dementia and with a Mini-Mental State Examination (MMSE) score >24 were included.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
The Barthel Index for Activities of Daily Living (ADL) | 24 hours
  ADL was evaluated on a scale of 100 points according to the patients' ability to feed themselves, bathe, perform personal hygiene, dress and undress, control bowel and bladder, use the toilet independently, use a wheelchair, mobility status, and ability to climb stairs.

SECONDARY OUTCOMES:
The Lawton-Brody Instrumental Activities of Daily Living (IADL) | 24 hours
  IADL consisted of eight sections, including the ability to use a telephone, shop, prepare meals, clean the house, do laundry, take medication, travel, and manage finances, and was evaluated on a scale of 17 points. Low scores were considered an indicator of dependence.
Walking speed | 2 minute
  For walking speed, the time to walk a 4.5-meter distance was measured.
Hand grip strength | 1 minute
  Hand grip strength of the dominant hand was measured twice with a Jamar dynamometer while sitting with the elbow flexed at 90 degrees, and the highest value was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Oztin, MD, Principal Investigator — Izmir Katip Celebi University, Ataturk Education And Research Hospital,

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fox C, Richardson K, Maidment ID, Savva GM, Matthews FE, Smithard D, Coulton S, Katona C, Boustani MA, Brayne C. Anticholinergic medication use and cognitive impairment in the older population: the medical research council cognitive function and ageing study. J Am Geriatr Soc. 2011 Aug;59(8):1477-83. doi: 10.1111/j.1532-5415.2011.03491.x. Epub 2011 Jun 24. PMID 21707557
- [Background] Lechevallier-Michel N, Molimard M, Dartigues JF, Fabrigoule C, Fourrier-Reglat A. Drugs with anticholinergic properties and cognitive performance in the elderly: results from the PAQUID Study. Br J Clin Pharmacol. 2005 Feb;59(2):143-51. doi: 10.1111/j.1365-2125.2004.02232.x. PMID 15676035
- [Result] Prasad S, Sung B, Aggarwal BB. Age-associated chronic diseases require age-old medicine: role of chronic inflammation. Prev Med. 2012 May;54 Suppl(Suppl):S29-37. doi: 10.1016/j.ypmed.2011.11.011. Epub 2011 Dec 9. PMID 22178471
- [Result] Jansen PA, Brouwers JR. Clinical pharmacology in old persons. Scientifica (Cairo). 2012;2012:723678. doi: 10.6064/2012/723678. Epub 2012 Jul 28. PMID 24278735